CLINICAL TRIAL: NCT00827658
Title: Ulnar Nerve Block for Procedural Anesthesia - Wrist Versus Palm
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Hamilton Health Sciences Corporation (Other)
Collaborators: McMaster University (Other)
Responsible Party: Sponsor
Organization: McMaster University (Other)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: McMaster 08-053
Record Dates: First submitted 2009-01-21; First posted 2009-01-23 (Estimated); Last update posted 2018-05-14 (Actual); Status verified 2018-05

CONDITIONS: Hand Surgery
Keywords: anesthesia, local; ulnar nerve; hand; surgery, plastic; blinded; randomized; prospective; local anesthesia; volar wrist block; hypothenar palm block; hand surgery

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hypothenar Palm block (Active Comparator): Hypothenar Palmar block group. Local anesthetic is placed at this location in this study group. The same local composition (Intervention) is used for both study groups. The trial is a comparison of location not the Intervention.
  Interventions: Procedure: Hypothenar Palm block
- Volar Wrist Block (Active Comparator): Volar Wrist block group. Local anesthetic is placed at this location in this study group. The same local composition (Intervention) is used for both study groups. The trial is a comparison of location not the Intervention.
  Interventions: Procedure: Volar Wrist Block

INTERVENTIONS:
Procedure: Volar Wrist Block — Injection medial to Flexor Carpi Ulnaris Tendon at volar proximal wrist crease
  Local Block - total 3 cc injection (1.5 cc 1% plain lidocaine and 1.5 cc of 0.25% bupivicaine)
  Arms: Volar Wrist Block
Procedure: Hypothenar Palm block — Injection at Hook of the Hamate on Palmar surface
  Local Block - total 3 cc injection (1.5 cc 1% plain lidocaine and 1.5 cc of 0.25% bupivicaine)
  Arms: Hypothenar Palm block

SUMMARY:
Ulnar nerve blockade is necessary for sensory anesthesia and analgesia in the hand during minor procedures. The course of the ulnar nerve in the forearm, wrist, and hand is predictable and has low variability. However even with known anatomic location and landmarks, ulnar nerve blocks at the wrist frequently are inadequate for procedural anesthesia. The antebrachial fascia at the wrist acts as a barrier to local infiltration. Since the fascia can not be visualized or palpated, it is commonly not penetrated, resulting in an inadequate block. Furthermore at the level of the wrist the ulnar artery lies in close proximity to the nerve and there is potential for arterial puncture while attempting injection for volar wrist block. The palmar ulnar nerve block is an injection distal to the hook of the hamate in the thenar eminence which avoids the ulnar artery and antebrachial fascia. This block has been used successfully for many years in clinical practice but has not been assessed or compared in a research study. The purpose of this study is to assess the validity of using a palmar ulnar nerve block for procedures in the hand as compared to the standard volar wrist ulnar nerve block.

ELIGIBILITY:
Inclusion Criteria:

* any individual who can give informed consent and is scheduled for elective hand procedures by the PI necessitating an Ulnar nerve block of the hand.

Exclusion Criteria:

* patients unable to give informed consent
* patients with previous or ongoing ulnar nerve deficits or neuropathy
* patients undergoing Guyon's canal decompression
* patients who can not comprehend or cooperate with assessment testing
* patients with abnormal two point discrimination (> 6 mm at the test location) prior to the nerve block

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2008-02; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Primary outcome is efficacy of sensory anesthesia and analgesia | 15-45 minutes

SECONDARY OUTCOMES:
Secondary outcome is patient perceived discomfort with block | 15-45 Minutes

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Martin, Principal Investigator — McMaster University
Locations (1):
- Hamilton General Hospital, Hamilton, Ontario, Canada